CLINICAL TRIAL: NCT05856916
Title: Creatine Supplementation for Improved Voice Performance in the Elderly
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Project is on indefinite hold due to a lack of funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-01536
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Presbyphonia
Keywords: creatine; presbyphonia; presbylarynx; vocal atrophy
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine Supplementation (Experimental): Participants randomized to receive creatine. Study participants will be asked to track their daily administration on a log provided by the study team.
  Interventions: Dietary Supplement: Creatine monohydrate
- Placebo (Placebo Comparator): Participants randomized to receive placebo. Study participants will be asked to track their daily administration on a log provided by the study team.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — Creatine monohydrate will be self-administered by an oral route at a dose of 5g/day in powdered form. Administration will begin on Study Day 1 and continue for 10 weeks.
  Other Names: Creapure
  Arms: Creatine Supplementation
Dietary Supplement: Placebo — Placebo (in the form of lactose) will be self-administered by an oral route at a dose of 5g/day in powdered form. Administration will begin on Study Day 1 and continue for 10 weeks.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine if creatine supplementation improves acoustic, auditory perceptual, physiologic, and patient-reported outcome measures in patients over 65 years of age. In the study, 20 participants will be enrolled and randomly assigned to receive either creatine or placebo.

DETAILED DESCRIPTION:
This will be a double-blinded, placebo-controlled interventional trial. Participants will be 65 years or older who present to the NYU voice center for voice complaints and desired voice therapy for improved vocal performance. Upon enrollment, participants will undergo evaluation for measures of vocal function (acoustic and aerodynamic measures of voice production), laryngeal physiology (electroglottography, videostroboscopy), and voice-associated quality of life (voice handicap index 10 , OMNI vocal effort scale, aging voice index). Participants will be randomized to receive either daily oral creatine supplementation or placebo. After 4 weeks, repeat measures will be taken. At this time, participants will initiate a standard-of-care course of voice therapy directed at improved vocal strength and endurance. The duration of therapy will be approximately 6 weeks. Participants will continue creatine supplementation or placebo through the course of therapy and repeat measures will be assessed at the conclusion of voice therapy. This will mark the end of the study period for each subject.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older
2. Desiring to participate in voice therapy

Exclusion Criteria:

1. Lesions or abnormalities of the larynx not attributable to normal aging
2. Pre-existing renal disease
3. Pre-existing liver disease
4. Congestive heart failure
5. Blood urea nitrogen (BUN), creatine, alanine transaminase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma-glutamyl transpeptidase (GGT) over reference range in the last 6 months
6. Concurrent medication associated with reduced renal clearance (e.g. Nonsteroidal Anti-inflammatory Drugs (NSAIDs), metformin)
7. History of prior vocal fold augmentation procedures
8. Cognitive disability
9. Unwillingness to participate in voice therapy

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Voice Handicap Index (VHI)-10 Scores | Baseline, Week 10
  10-item questionnaire assessing a patient's perception of impairment or handicap due to a voice problem. Items are ranked on a scale ranging from 0 to 4, where 0 = Never and 4 = Always. The total score ranges from 0-40; higher scores indicate greater impairment or handicap due to a voice problem.
Average Expert Rating of Change in Mucosal Wave | Week 10
  Videostroboscopic clips will be collected during clinical visits (baseline and Week 10). The clips will be sent to 6 expert reviewers, who will rate change in mucosal wave on a relative 3-point scale (1 = worse, 2 = same, 3 = better).
Average Expert Rating of Change in Vocal Fold Atrophy | Week 10
  Videostroboscopic clips will be collected during clinical visits (baseline and Week 10). The clips will be sent to 6 expert reviewers, who will rate change in vocal fold atrophy on a relative 3-point scale (1 = worse, 2 = same, 3 = better).
Average Expert Rating of Change in Glottal Closure | Week 10
  Videostroboscopic clips will be collected during clinical visits (baseline and Week 10). The clips will be sent to 6 expert reviewers, who will rate change in glottal closure on a relative 3-point scale (1 = worse, 2 = same, 3 = better).
Average Phonatory Pressure during Aerodynamic Analysis of Voice | Up to Week 10
  Patients are instructed to produce five productions of /pa/ at their most comfortable pitch and loudness at a rate of approximately 1.5 syllables per second. The middle three productions will be analyzed to determine the average phonatory pressure.
Average Decibel (dB) Output during Aerodynamic Analysis of Voice | Up to Week 10
  Patients are instructed to produce five productions of /pa/ at their most comfortable pitch and loudness at a rate of approximately 1.5 syllables per second. The middle three productions will be analyzed to determine the average dB output.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Johnson, Principal Investigator — Aaron.Johnson@nyulangone.org
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a single institution study and all patient data will be limited to the primary research team